CLINICAL TRIAL: NCT07161401
Title: Sagittal Skeletal Malocclusions and Sleep Quality in Children Without Orofacial Dysfunction
Brief Title: Sagittal Malocclusion and Sleep Quality in Children
Status: Completed | Type: Observational
Sponsor: Serap Titiz Yurdakal (Other)
Responsible Party: Sponsor-Investigator, Serap Titiz Yurdakal, Associate Professor of Orthodontics, Faculty of Dentistry, Dokuz Eylül University, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Other Study IDs: 06-06-11
Record Dates: First submitted 2025-08-30; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Sleep Quality
Keywords: Pediatric sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Skeletal Class I: Participants with skeletal Class I malocclusion based on ANB angle.
  Interventions: Other: Observational assessment
- Group 2: Skeletal Class II: Participants with skeletal Class II malocclusion based on ANB angle.
  Interventions: Other: Observational assessment
- Group 3: Skeletal Class III: Participants with skeletal Class III malocclusion based on ANB angle.
  Interventions: Other: Observational assessment

INTERVENTIONS:
Other: Observational assessment — Evaluation of sleep quality using the Children's Sleep Habits Questionnaire (CSHQ) and cephalometric analysis of mandibular position (SNB), vertical dimensions (SNGoGn, FMA), and upper airway measurements. No active intervention was performed.

SUMMARY:
This observational cross-sectional study evaluated the impact of sagittal skeletal malocclusions on sleep quality in children without orofacial functional disorders. A total of 164 children aged 7-13 years were assessed. Sleep quality was measured using the Children's Sleep Habits Questionnaire (CSHQ), and participants were classified as skeletal Class I, II, or III based on cephalometric analyses. Comparisons were made between skeletal groups regarding CSHQ scores, mandibular and vertical skeletal measurements, and upper airway dimensions. The aim was to determine whether skeletal discrepancies independently influence pediatric sleep quality in the absence of functional impairments.

DETAILED DESCRIPTION:
This observational cross-sectional study investigated the potential impact of sagittal skeletal malocclusions on sleep quality in children without orofacial functional disorders. Sleep and craniofacial growth are closely related, and functional disturbances such as atypical swallowing or thumb-sucking are known to influence both airway patency and sleep. To isolate the independent role of skeletal discrepancies, children with orofacial dysfunction were excluded. A total of 164 children aged 7-13 years were evaluated. Sleep quality was measured using the Children's Sleep Habits Questionnaire (CSHQ). Based on cephalometric analysis, participants were classified into skeletal Class I, II, or III according to the ANB angle. Additional cephalometric parameters, including mandibular position (SNB), vertical skeletal dimensions (SNGoGn and FMA angles), and two-dimensional upper airway dimensions, were recorded. For each skeletal group, comparisons were made regarding demographic data, sleep scores, and craniofacial measurements. Correlations between CSHQ scores and cephalometric values were further analyzed separately in male and female patients. The results showed significant differences in mandibular positioning across skeletal groups, with males in Class II presenting higher vertical values than those in Class I or III. However, no significant differences were found between skeletal groups in terms of sleep quality or airway dimensions, and no correlation was observed between sleep quality scores and skeletal measurements in either sex. In conclusion, the findings suggest that, in the absence of orofacial functional disorders, sagittal skeletal malocclusions alone may not significantly affect pediatric sleep quality. This study highlights the importance of differentiating skeletal anomalies from functional disturbances when investigating the complex relationship between craniofacial development and sleep in children.

ELIGIBILITY:
Inclusion Criteria:

Children aged 7-13 years

Presence of skeletal Class I, II, or III malocclusion (based on ANB angle)

Written informed parental consent

Exclusion Criteria:

Presence of systemic diseases

Current use of medications such as anticonvulsants, immunosuppressants, or calcium channel blockers

Exposure to stressful life events within the past month

Presence of deleterious oral habits (e.g., thumb sucking, mouth breathing, infantile swallowing)

Signs of tonsillar hypertrophy, nasal deviation, nasal polyps, or adenoid vegetation

Diagnosis of sleep-disordered breathing (SDB)

History of orofacial surgery or orthodontic treatment

Presence of craniofacial anomalies (e.g., cleft lip/palate, syndromes)

Ages: 7 Days to 13 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population consisted of children aged 7-13 years presenting with skeletal Class I, II, or III malocclusion. Only patients without systemic diseases, orofacial functional disorders, previous orthodontic treatment, or craniofacial anomalies were included
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Sleep Quality (CSHQ Score) | At baseline (single assessment)
  Sleep quality was assessed using the Children's Sleep Habits Questionnaire (CSHQ), a validated parent-reported tool. Higher total scores indicate poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Uşak University, Faculty of Dentistry, Department of Orthodontics, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data (IPD) will be available from the corresponding author upon reasonable request, after publication of the study results.